CLINICAL TRIAL: NCT00645983
Title: Chamomile Therapy for Generalized Anxiety Disorder
Brief Title: Chamomile Therapy for Generalized Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Jay D. Amsterdam, M.D., Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AT001916 (NIH); R21AT001916 (NIH)
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Generalized Anxiety Disorder
Keywords: Chamomile; Anxiety; Complementary and Alternative Medicine
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Chamomile extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Chamomile Extract
  Interventions: Dietary Supplement: Chamomile Extract
- 2 (Placebo Comparator): Anxiolytic Therapy
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Chamomile Extract — 220 mg - 1100 mg daily
  Arms: 1
Other: Placebo — 1 to 5 capsules daily
  Arms: 2

SUMMARY:
This study will determine the effectiveness of chamomile extract for treating generalized anxiety disorder.

Study hypotheses: 1)Chamomile extract will have a superior anti-anxiety effect compared to placebo. 2)Chamomile will have a comparable safety profile to that of placebo.

DETAILED DESCRIPTION:
We propose to investigate the anti-anxiety activity of Chamomile. Among the many uses of Chamomile, its use as an anti-anxiety herb is universal. Despite its widespread use and acceptance, there have been no studies evaluating the safety and anti-anxiety efficacy of Chamomile in human subjects. Given this lack of controlled clinical data, we propose a pilot study of Chamomile safety and efficacy in mild anxiety, and propose using the data as a basis for statistically powering a future R01 application. We will ask: Is Chamomile a safe and effective alternative treatment for Generalized Anxiety Disorder (GAD)? To do this, 60 patients with a diagnosis of mild to moderate GAD will receive double-blind treatment for 8 weeks with either (i) Chamomile extract, or (ii) placebo. We hypothesize that Chamomile will have a superior anti-anxiety efficacy compared to placebo, and a comparable safety profile to placebo.

ELIGIBILITY:
Inclusion Criteria:

Men and women > 18 years of age (all races and ethnicity)

Meet DSM IV criteria for GAD

Mild to moderate symptom severity

HAM-A score > 8

Not receiving anti-anxiety medication (e.g., benzodiazepine, venlafaxine, buspirone, or SSRI)

Able to understand and provide signed informed consent

Able to participate in a 8-week study

Exclusion Criteria:

Patients < 18 years old

Current DSM IV Axis I diagnosis of Major Depressive Disorder, Bipolar Disorder, Panic Disorder (with or without agoraphobia), Specific Phobia Disorder, Obsessive-Compulsive Disorder, Posttraumatic Stress Disorder, Acute Stress Disorder, Substance-Induced Anxiety Disorder, Schizophrenia, Other psychotic disorders, Current alcohol or drug abuse, Alcohol or drug dependence within 3 months, [NB: Patients with co-morbid DSM IV Axis I Depressive Disorders NOS (e.g., minor depressive disorder, premenstrual dysphoric disorder, and recurrent brief depressive disorder will not be excluded)]

Unstable medical condition (e.g., hypothyroidism, hypertension, myocardial infarction within 1 month, neoplastic condition)

Allergy to Chamomile preparation

Allergy to plants of the asteraceae family (e.g., ragweed, asters, chrysanthemum)

Allergy to mugwort, RAST, or birch tree pollen

Concurrent tranquilizer, antidepressant or mood stabilizer therapy

Concurrent use of over-the-counter anti-anxiety and/or antidepressant preparations (e.g., Chamomile, St. John's Wort, Kava kava)

Women of child-bearing potential not willing to employ a medically proven form of contraception (e.g., condoms, oral contraceptives, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Score on Hamilton Anxiety Rating Scale | 8 Weeks

SECONDARY OUTCOMES:
Beck Anxiety Index Rating | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jay D. Amsterdam, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Depression Research Unit, Universityof Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Amsterdam JD, Li Y, Soeller I, Rockwell K, Mao JJ, Shults J. A randomized, double-blind, placebo-controlled trial of oral Matricaria recutita (chamomile) extract therapy for generalized anxiety disorder. J Clin Psychopharmacol. 2009 Aug;29(4):378-82. doi: 10.1097/JCP.0b013e3181ac935c. PMID 19593179